CLINICAL TRIAL: NCT00094705
Title: Phase 1 Study of the Safety and Immunogenicity of rDEN2/4delta30(ME), a Live Attenuated Virus Vaccine Candidate for the Prevention of Dengue Serotype 2
Brief Title: Safety of and Immune Response to a Dengue Virus Vaccine (rDEN2/4delta30[ME]) in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Johns Hopkins Bloomberg School of Public Health (Other)
Responsible Party: Anna Durbin, MD, Center for Immunization Research, Johns Hopkins School of Public Health
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CIR 189; H.22.03.09.26.A2
Record Dates: First submitted 2004-10-21; First posted 2004-10-22 (Estimated); Last update posted 2008-01-21 (Estimated); Status verified 2008-01

CONDITIONS: Dengue Fever
Keywords: Dengue Vaccine; Dengue Virus; Dengue Hemorrhagic Fever; Dengue Shock Syndrome
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): One subcutaneous vaccination with a 10^3 PFU dose of rDEN2/4delta30(ME) vaccine given in the deltoid region of either arm.
  Interventions: Biological: rDEN2/4delta30(ME) Vaccine
- 2 (Experimental): One subcutaneous vaccination with a 10^5 PFU dose of rDEN2/4delta30(ME) vaccine given in the deltoid region of either arm.
  Interventions: Biological: rDEN2/4delta30(ME) Vaccine
- 3 (Placebo Comparator): One subcutaneous vaccination with a placebo vaccine given in the deltoid region of either arm.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: rDEN2/4delta30(ME) Vaccine — Live attenuated rDEN2/4delta30(ME) vaccine (one of two doses)
  Arms: 1; 2
Biological: Placebo — Placebo for rDEN2/4delta30(ME) vaccine
  Arms: 3

SUMMARY:
Dengue fever, which is caused by dengue viruses, is a major health problem in tropical and subtropical regions of the world. The purpose of this study is to test the safety of and immune response to a new dengue virus vaccine in healthy adults.

DETAILED DESCRIPTION:
Dengue viruses cause dengue fever, as well as the more severe dengue hemorrhagic fever/shock syndrome. More than 2 billion people living in tropical and subtropical regions of the world are at risk of dengue virus infection, which is the leading cause of hospitalization and death in children in several tropical Asian countries. This study will evaluate the safety and immunogenicity of a live attenuated dengue virus vaccine called rDEN2/4delta30(ME), which is derived from the DEN2 and DEN4 serotypes.

This study will last 180 days. Participants in Cohort 1 will be randomly assigned to receive rDEN2/4delta30(ME) or placebo at study entry. Cohort 2 will begin only after safety review of all participants in Cohort 1. Participants in Cohort 2 will receive a higher dose of rDEN2/4delta30(ME) or placebo.

After vaccination, participants will be observed for at least 30 minutes for immediate adverse reactions. Participants will also be asked to monitor their temperature every day for 16 days. Study visits will occur every other day after vaccination until Day 16, followed by 4 additional visits at selected days through Day 180. Blood collection and a targeted physical exam will occur at each study visit. Some participants will be asked to undergo a skin biopsy or additional blood collection at selected visits.

ELIGIBILITY:
Inclusion Criteria:

* Willing to be followed for the duration of the study
* Willing to use acceptable methods of contraception
* Good general health

Exclusion Criteria:

* Clinically significant neurologic, cardiac, pulmonary, hepatic, rheumatologic, autoimmune, or renal disease
* Behavioral, cognitive, or psychiatric disease that, in the opinion of the investigator, affects the ability of the volunteer to understand and cooperate with the study
* Hematologic disease
* Alcohol or drug abuse within 12 months prior to study entry
* History of severe allergic reaction or anaphylaxis
* Emergency room visit or hospitalization for severe asthma within 6 months prior to study entry
* HIV-1 infected
* Hepatitis C virus infected
* Hepatitis B surface antigen positive
* Known immunodeficiency syndrome
* Use of corticosteroids or immunosuppressive drugs within 30 days prior to study entry. Participants who have used topical or nasal corticosteroids are not excluded.
* Live vaccine within 4 weeks prior to study entry
* Killed vaccine within 2 weeks prior to study entry
* Blood products within 6 months prior to study entry
* Participation in another investigational vaccine or drug trial within 60 days of starting this study, or while this trial is ongoing
* Previously received a licensed or experimental yellow fever or dengue vaccine
* Surgical removal of spleen
* History of dengue virus infection or other flavivirus infection (e.g., yellow fever virus, St. Louis encephalitis, West Nile virus, Japanese encephalitis virus)
* Other condition that, in the opinion of the investigator, would affect the participant's participation in the study
* Plan to travel to an area where dengue infection is common
* Pregnancy or breastfeeding

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2005-01; Primary Completion 2006-04 (Actual); Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of vaccine-related adverse effects for each dose graded by severity | Throughout study
Amount of dengue 2 neutralizing antibody induced by the vaccine | At Day 42

SECONDARY OUTCOMES:
To assess the durability of the antibody response out to Day 180 | Throughout study
To assess the frequency, quantity, and duration of viremia in each dose cohort studied | Throughout study
To determine the number of vaccinees infected with rDEN2/4delta30(ME) | Throughout study
To compare the T cell mediated immune response against dengue viruses of those volunteers infected with the rDEN2/4delta30(ME) vaccine virus with that of uninfected volunteers and placebo recipients | Throughout study
If both doses of vaccine are administered, to compare the infectivity rates, safety, and immunogenicity between dose groups | At study completion
To evaluate the immunopathological mechanism of vaccine-associated rash in those volunteers who are willing to undergo skin biopsy | Throughout study

CONTACTS AND LOCATIONS:
Overall Officials: Anna Durbin, MD, Principal Investigator — Center for Immunization Research, Johns Hopkins School of Public Health
Locations (1):
- Johns Hopkins School of Public Health, Baltimore, Maryland, United States

REFERENCES:
- [Background] Edelman R. Dengue and dengue vaccines. J Infect Dis. 2005 Mar 1;191(5):650-3. doi: 10.1086/427784. Epub 2005 Jan 27. No abstract available. PMID 15688277
- [Background] Guzman MG, Mune M, Kouri G. Dengue vaccine: priorities and progress. Expert Rev Anti Infect Ther. 2004 Dec;2(6):895-911. doi: 10.1586/14789072.2.6.895. PMID 15566333
- [Background] Sabchareon A, Lang J, Chanthavanich P, Yoksan S, Forrat R, Attanath P, Sirivichayakul C, Pengsaa K, Pojjaroen-Anant C, Chokejindachai W, Jagsudee A, Saluzzo JF, Bhamarapravati N. Safety and immunogenicity of tetravalent live-attenuated dengue vaccines in Thai adult volunteers: role of serotype concentration, ratio, and multiple doses. Am J Trop Med Hyg. 2002 Mar;66(3):264-72. doi: 10.4269/ajtmh.2002.66.264. PMID 12139219
- [Background] Sun W, Edelman R, Kanesa-Thasan N, Eckels KH, Putnak JR, King AD, Houng HS, Tang D, Scherer JM, Hoke CH Jr, Innis BL. Vaccination of human volunteers with monovalent and tetravalent live-attenuated dengue vaccine candidates. Am J Trop Med Hyg. 2003 Dec;69(6 Suppl):24-31. doi: 10.4269/ajtmh.2003.69.6_suppl.0690024. PMID 14740952
- [Background] Whitehead SS, Hanley KA, Blaney JE Jr, Gilmore LE, Elkins WR, Murphy BR. Substitution of the structural genes of dengue virus type 4 with those of type 2 results in chimeric vaccine candidates which are attenuated for mosquitoes, mice, and rhesus monkeys. Vaccine. 2003 Oct 1;21(27-30):4307-16. doi: 10.1016/s0264-410x(03)00488-2. PMID 14505913